CLINICAL TRIAL: NCT03446924
Title: Determining the Muscle Anabolic Properties of Phosphatidic Acid in Ageing.
Brief Title: Determining the Muscle Anabolic Properties of Phosphatidic Acid.
Acronym: PA-AGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RG_14-192
Record Dates: First submitted 2018-02-15; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Sarcopenia
Keywords: Nutraceuticals; Muscle anabolism; Ageing
MeSH Terms: conditions — Sarcopenia | interventions — Phosphatidic Acids; Flour

STUDY DESIGN:
Intervention Model Description: Parallel-designed study in which participants will be randomized to receive phosphatidic acid or placebo treatment. A parallel design was chosen due to the number of invasive muscle biopsies performed during each experimental trial.
Who Masked: Participant, Investigator
Masking Description: An individual with no direct study involvement will administer treatments in a double-blind manner. Investigators will be un-blinded to treatment arms upon completion of data analysis.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): The control group will be given a single dose of 1.5 g rice flour in capsule form (250 mg / capsule). The gelatine capsules (MyProtein, Northwich, UK) used are identical to those used in the treatment group. Capsules are prepared by the investigatory team using good hygiene practice in the research kitchen of the School of Sport, Exercise and Rehabilitation (University of Birmingham).
  Interventions: Dietary Supplement: Rice flour
- Treatment (Active Comparator): The treatment group will be given a single dose of 1.5g phosphatidic acid in capsule form (250 mg / capsule). Capsules are prepared by the investigatory team using good hygiene practice in the research kitchen of the School of Sport, Exercise and Rehabilitation (University of Birmingham).
  PA is considered a dietary supplement ingredient according to the US FDA. The source of PA will be a commercial available soy-derived PA (Mediator®, Chemi Nutra, White Bear Lake, MN). The safety of Mediator® Soy-PA has been thoroughly demonstrated in humans. Mediator® Soy-PA does not contain any compounds with narcotic, psychotropic or pharmaceutical effects and is in compliance with banned substances requirements as espoused by the World Anti-Doping Agency. Mediator® Soy-PA is not a medicinal product.
  Interventions: Dietary Supplement: Phosphatidic Acid

INTERVENTIONS:
Dietary Supplement: Phosphatidic Acid — To be administered a single dose of 1.5 g phosphatidic acid in capsule form (250 mg / capsule).
  Arms: Treatment
Dietary Supplement: Rice flour — Rice flour placebo to be administered a single dose of 1.5 g in capsule form (250 mg / capsule).
  Arms: Control

SUMMARY:
Ageing is characterized by a loss of muscle mass that is detrimental for physical function and metabolic health and increases the risk of mortality. The loss of muscle protein mass with ageing is characterized by a blunted muscle anabolic response to nutrition and exercise. Thus, interventions to counteract muscle anabolic blunting in old age might assist in the long-term maintenance of muscle mass.

Phosphatidic acid (hereafter defined as 'PA') is a novel nutrient compound that has been suggested to play an important role in muscle growth. Oral consumption of PA may amplify the signalling response to nutrition and exercise and restore muscle anabolic sensitivity in older adults. In order for PA to be 'clinically' applied as a means to mitigate muscle loss in aged populations, we must first understand the efficacy and mechanisms underlying the anabolic properties of this compound, which have yet to be defined in man. The proposed pilot study is needed to investigate the acute muscle metabolic properties of oral PA supplementation in older individuals.

Sixteen healthy (non-obese, non-diabetic, non-smokers) older males aged 65-75 yrs will initially complete a lower-limb strength assessment and undergo a body composition scan. Between 4-14 days after these initial assessments, participants will be assigned to co-ingest 1.5g of either phosphatidic acid (N= 8; PA) or a non-caloric placebo (N=8; PL) after following a bout of moderate intensity, single leg resistance exercise. A stable isotope infusion will be combined with serial muscle biopsies from the thigh of each leg to determine the measure rates of muscle protein synthesis in the fasted state and in the 'early' and 'late' phase of feeding-only and exercise-plus-feeding.

DETAILED DESCRIPTION:
The investigators will recruit 16 healthy (non-obese, non-diabetic, non-smokers) elderly men aged 65-80 yrs to complete a double-blinded, parallel designed study, in which they will be randomly assigned to a phosphatidic acid (N= 8; PA) or placebo (N=8; PL) treatment group, matched closely for anthropometric characteristics. Participants will be recreationally active, but not involved in structured exercise training. All study procedures will be clearly explained and written consent obtained prior to study participation.

Preliminary assessments Following explanation of the study and the acquisition of informed consent, participants will report to our laboratory at 0800 in an overnight fasted-state and having refrained from strenuous physical activity for >24 hrs. Participants will be weighed on a digital scale to the nearest 0.1 kg in light clothing. A dual x-ray absorptiometry (DXA) scan will be conducted to determine body composition (fat and fat-free mass). Following DXA scanning, single-leg one repetition maximum strength (1RM) will be determined for knee extension and leg press exercise machines. Selection of the limb to be exercised (dominant or non-dominant) will be randomized.

Experimental trials Between 4 and 14 days after the preliminary assessments, participants will report to the laboratory at ∼0700 following an overnight fast, having refrained from strenuous physical activity for 72 hrs previously. A catheter will be inserted into a forearm vein of both arms for frequent blood sampling (∼80mL in total) and a continuous infusion of a stable isotope amino acid tracer (L- [ring] 13C6 phenylalanine). Participants will remain in a supine position throughout the trial with the exception of the exercise bout. After 150 min of steady-state tracer infusion a muscle biopsy will be obtained from the vastus lateralis quadriceps muscle of a randomly selected leg under local anesthesia (1% lidocaine) using the Bergström biopsy needle technique. Thereafter, participants will perform a bout of single-leg resistance exercise on the opposite leg. Exercise will consist of 6 sets of knee extension resistance exercise at 75% of the pre-determined 1RM; a protocol designed to elicit 8-12 repetitions per set prior to the onset of volitional fatigue. Immediately after exercise, participants will ingest 750mg of PA or a placebo (both in non-identifiable capsule form) with water and a further 750mg of PA or placebo at 60 mins post-exercise. Thereafter, participants will lie in a supine position for the remainder of the trial. An individual with no direct study involvement will administer treatments in a double-blind manner. Investigators will be un-blinded to treatment arms upon completion of data analysis. At 150 and 300 min following treatment consumption muscle biopsies will be obtained from both legs. Thus, a total of 5 invasive muscle biopsies will be obtained during the trial, which precludes the use of a crossover design in older individuals. Each biopsy will be obtained from a separate incision spaced ∼3cm apart. This model of study design will permit us determine rates of muscle protein synthesis in the postabsorptive state and over the early (0-2.5 h), late (2.5-5 h) and aggregate (0-5 h) time-course.

Data Analyses To calculate muscle protein synthesis, the investigators will adopt sophisticated mass spectrometry techniques to determine isotopic tracer enrichment in biopsy-isolated muscle proteins and plasma. Intramuscular "anabolic signals" (in the mechanistic target of rapamycin pathway, a key regulator of cell size) will be determined via Western Blot (a technique to detect the content of specific phospho-proteins). Plasma insulin concentrations will be measured by immunoassay and plasma lipid profiles by Gas Chromatography Mass Spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Be a non-smoking male between 65 and 80 years.
* Have a BMI between 18 and 25 kg/m2.
* Be in good general health: no cardiovascular or metabolic diseases.

Exclusion Criteria:

* Health problems such as: heart disease, rheumatoid arthritis, uncontrolled hypertension, poor lung function, or any health condition that might put you at risk when participating in this study.
* Generalised neuromuscular disease (such as Parkinson's disease or motorneurone disease).
* Failure to obtain clearance for exercise participation from your GP or negative advice given by your GP concerning exercise participation.
* Involvement in regular structured resistance exercise training at the time of the study.
* Consumption of any analgesic drugs, anti-inflammatory drugs, or medication that is known to affect protein metabolism (beta-blockers, corticosteroids, NSAIDs).
* Participants who have undergone muscle biopsy testing or isotope infusion procedures within the last 5 years.

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Myofibrillar protein synthesis in response to oral phosphatidic acid or placebo ingestion alone or in combination with resistance exercise | The change in myofibrillar protein synthesis after treatment ingestion will be determined over 0-to-2.5 hours and 2.5-to-5 hours post-ingestion in rested and exercised legs
  Myofibrillar protein synthesis will be determined via mass spectrometry to assess stable isotope enrichment of 13C6 phenylalanine isotope in the myofibrillar protein fraction of biopsy tissue. The standard precursor-product calculations will be applied, using plasma isotope enrichment as the precursor.

SECONDARY OUTCOMES:
Anabolic and proteolytic signalling phosphorylation | The change in signaling protein phosphorylation from rest will be measured at 2.5 and 5 h after treatment ingestion in rested and exercised legs
  Phosphorylation of key anabolic and proteolytic signalling intermediates that modulate myofibrillar protein synthesis will be determined via western blot technique

CONTACTS AND LOCATIONS:
Locations (1):
- University of Birmingham, School of Sport, Exercise and Rehabilitation Sciences, Edgbaston, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smeuninx B, Nishimura Y, McKendry J, Limb M, Smith K, Atherton PJ, Breen L. The effect of acute oral phosphatidic acid ingestion on myofibrillar protein synthesis and intracellular signaling in older males. Clin Nutr. 2019 Jun;38(3):1423-1432. doi: 10.1016/j.clnu.2018.06.963. Epub 2018 Jun 21. PMID 29970319